CLINICAL TRIAL: NCT06405295
Title: A Multicentre Prospective Cohort Study: Intensive Adjuvant Therapy for TNBC with BRCA Gene Mutation
Brief Title: Intensive Adjuvant Therapy for TNBC with BRCA Gene Mutation
Status: Enrolling by invitation | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, PENG YUAN, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC3896
Record Dates: First submitted 2024-05-04; First posted 2024-05-08 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-05

CONDITIONS: Breast Carcinoma; BRCA Mutation; Adjuvant Drug Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — BRCA gene testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Capecitabine
  Interventions: Other: no intervention
- Olaparib
  Interventions: Other: no intervention
- Capecitabine and Olaparib
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — Observation of the prognosis of patients with different standard treatment protocols in the clinic without intervention

SUMMARY:
Evaluation of the efficacy and safety of different adjuvant intensification regimens in early-stage BRCA1/2 mutant triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* ECOG score 0-1
* TNBC
* BRCA1/2 mutation
* No distant metastases assessed by imaging after surgical treatment
* Breast cancer that is non-pCR after neoadjuvant therapy, or postoperative pathology suggestive of ≥pT2, or ≥pN1
* Have completed postoperative adjuvant chemotherapy and/or radiotherapy
* No major organ dysfunction

Exclusion Criteria:

* Patients who are unable to take oral medication, or who refuse this medication regimen
* Already enrolled in another study, or less than or equal to 4 weeks from discontinuation of another medication
* Presence of severe dysfunction of vital organs
* Patients with other malignancies (with the exception of cured non-melanoma skin cancers, carcinoma in situ of the cervix and other tumours that have been cured for at least 5 years)
* Acute infectious disease or active chronic infectious disease
* History of uncontrolled epilepsy, central nervous system disease or mental disorder

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early-stage triple-negative breast cancer with BRCA1/2 mutations treated at multiple hospitals in China with postoperative sequential treatment with capecitabine or olaparib or a combination of both drugs
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
iDFS% | 3 years

SECONDARY OUTCOMES:
DRFS% | 3 years
OS% | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, Principal Investigator
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No